CLINICAL TRIAL: NCT02517619
Title: A Prospective, Multi-Center, Randomized, Double-Masked, Positive Controlled, Phase 3 Clinical Trial Designed to Evaluate the Safety and Efficacy of Iontophoretic Dexamethasone Phosphate Ophthalmic Solution Compared to Prednisolone Acetate Ophthalmic Suspension (1%) in Patients With Non-Infectious Anterior Segment Uveitis
Brief Title: Safety and Efficacy of Iontophoretic Dexamethasone Phosphate Ophthalmic Solution in Non-Infectious Anterior Uveitis
Acronym: EGP-437-006
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eyegate Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EGP-437-006
Record Dates: First submitted 2015-08-05; First posted 2015-08-07 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Anterior Uveitis
Keywords: Iontophoresis; Ophthalmology; Non-Infectious Anterior Segment Uveitis
MeSH Terms: conditions — Uveitis, Anterior | interventions — prednylidene

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone Phosphate Ophthalmic Solution (Experimental): Dexamethasone phosphate ophthalmic solution (40 mg/mL)
  Interventions: Drug: Dexamethasone Phosphate Ophthalmic Solution
- Prednisolone Acetate Ophthalmic (1%) (Active Comparator): Prednisolone Acetate Ophthalmic (1%)
  Interventions: Drug: Prednisolone Acetate Ophthalmic (1%)

INTERVENTIONS:
Drug: Dexamethasone Phosphate Ophthalmic Solution — 40 mg/mL
  Other Names: EGP-437
  Arms: Dexamethasone Phosphate Ophthalmic Solution
Drug: Prednisolone Acetate Ophthalmic (1%) — Prednisolone Acetate (1%)
  Other Names: Pred Acetate (1%)
  Arms: Prednisolone Acetate Ophthalmic (1%)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ocular iontophoresis with dexamethasone phosphate ophthalmic solution EGP-437 using the EyeGate® II Drug Delivery System (EGDS) compared to prednisolone acetate ophthalmic suspension (1%) in patients with non-infectious anterior segment uveitis.

DETAILED DESCRIPTION:
This will be a Phase 3, randomized, double-masked, parallel arm, positive-controlled non-inferiority study, in which up to 250 subjects (approximately 125 subjects per treatment arm) will be enrolled at up to 60 clinical sites. Patients with non-infectious anterior segment uveitis who are interested in participating in the study will be provided an informed consent form prior to screening. Screening/Baseline procedures which include BCVA, slit lamp examination, fundus exam, IOP by tonometry will be used to determine eligibility.

ELIGIBILITY:
Inclusion Criteria:

1. Age 12 to 85 years with a diagnosis of non-infectious anterior segment uveitis defined as an AC cell count of ≥ 11 cells
2. Receive, understand, and sign a copy of the written informed consent form
3. Be able to return for all study visits and willing to comply with all study-related instructions

Exclusion Criteria:

Ages: 12 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2016-01-16 (Actual); Primary Completion 2018-04-20 (Actual); Study Completion 2018-05-29 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with an AC cell count of zero at Day 14 | Day 14 ± 2 days

CONTACTS AND LOCATIONS:
Overall Officials: John D. Sheppard, M.D., Principal Investigator — Study Principal Investigator
Locations (1):
- Virginia Eye Consultants, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes